CLINICAL TRIAL: NCT04736511
Title: Study of the Influence of Proprioceptive Reweighting Ability on the Lower-extremity Biomechanics During Functional Tasks and Unplanned Sidestep Cutting Manoeuvre
Brief Title: Influence of Proprioceptive Reweighting Ability on Lower-limb Biomechanics During Functional Tasks
Acronym: NEURIBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC20.0288 NEURIBIO
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2022-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: proprioceptive reweighting ability; sidestep cutting manoeuvre; handball
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Mono-centric comparative cross-sectional observational study with minimal risks and constraints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other): Handball players
  Interventions: Other: Star Excursion Balance Test; Other: Single leg Drop Vertical Jump; Other: Unplanned sidestep cutting manoeuvre; Other: Tendon vibration

INTERVENTIONS:
Other: Star Excursion Balance Test — The subject will be in unipodal support (only one foot on the ground) on the tested lower limb in the center of the platform. Three lines forming a "Y" will be arranged according to the lower limb in charge in three directions : anterior (ANT), posteromedial (PM) and posterolateral (PL). The goal is then to reach the longest distance possible in all three directions with the tip of the foot in relief before returning to the starting position. The subject will have 4 training trials per direction on each lower limb then 3 trials will be recorded in order to keep the average.
  Other Names: SEBT
Other: Single leg Drop Vertical Jump — The subject will drop from a step and land on one leg, then jump as high as possible and stabilize again on the same leg. The height of the step is 30 cm. The subject will perform 3 consecutive jumps in the strictest respect of the instructions: drop to the level of the mark on the ground and bounce as high as possible while spending a minimum of time on the ground. The subject must stabilize for 3 seconds during the second contact with the ground so that the instructions and measurements are reproducible.
  Other Names: SDVJ
Other: Unplanned sidestep cutting manoeuvre — The objective is to create an unanticipated playing situation, close to the daily actions of the subjects in the practice of handball. The subject will make sidestep cutting manœuvre in front of an opponent simulated by a dummy used during usual training.
  The subject will sprint in a straight line and then at the force platform will make a rapid change of direction on the side of his shooting arm or will continue his run in a straight line. A light signal randomly will indicate to the player the direction in which he must carry out his manoeuvre. A computer reconstruction of the kinematics and dynamics (knee moment) will be performed.
  Other Names: Unplanned change of direction
Other: Tendon vibration — The subject will be asked to stand, motionless in bipodal (both feet on the ground) support on a stable and unstable ground (foam). A tendon vibration (80Hz) will be randomly applied to the subject in the Achilles tendons or paravertebral muscles. This vibration will cause an alteration of proprioceptive information in the vibrated area leading to a disruption of postural balance. Thus, according to the amount of displacement of the center of pressure (CoP), the proprioceptive weighting ratio (dRPW) is calculated to deduce therefrom the weight assigned by the CNS to the various proprioceptive inputs during the postural task.

SUMMARY:
Anterior cruciate ligament (ACL) injuries are frequent in handball especially among young players. Recent investigations highlighted the implication of the central nervous system as a potential risk factor for ACL rupture.

The ability to dynamically reweight proprioceptive signals according to postural conditions is crucial for balance control.

The aim of this study is therefore to investigate the influence of proprioceptive reweighting on biomechanical determinants of ACL loads during functional tasks and unplanned side cutting manoeuvers.

DETAILED DESCRIPTION:
Team Handball is a traumatic sport, especially regarding anterior cruciate ligament (ACL) injuries. Young females are more vulnerable as they are 3 to 5 times more likely to sustain an ACL rupture compare to males.

Several anatomical, biomechanical and sensorimotor risk factors have been clearly identified, however the implication of the central nervous system was recently highlighted. Indeed, it has been shown that individuals who will suffer of ACL ruptures exhibited a decreased functional connectivity between brain regions responsible for postural control and sensorimotor processing. Due to the unanticipated situations that occurred during game situations, the role of the brain (i.e neural control) is now advocated to explain sensorimotor errors leading to injuries during complex tasks such as faking an opponent. Muscle vibration is a reliable tool to assess proprioceptive integration during postural control. The ability to shift from one proprioceptive cue to another when postural conditions are changing is crucial. This dynamic reweighting process allow to obtain an optimal postural control. However, recent investigations revealed that this process is altered among symptomatic populations, elderly patients or even under fatigue conditions. More precisely, some individuals seem able to shift proprioceptive reliance while other doesn't. To our knowledge, no studies have investigated the link between proprioceptive reweighting and biomechanical determinants of ACL loads during functional tasks. Thus, the aim of this study is to compare lower-limb biomechanics during unanticipated side cutting manoeuvres and single leg drop vertical jump among young handball players according to their ability to reweight proprioceptive signals.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 15 to 25 years
* Intensive training handball practice for at least two years, mastering the technical gesture of unplanned sidestep cutting manoeuvre
* Training volume of 5 hours minimum per week
* Signature of the consent (participants and parents for minors)

Exclusion Criteria:

* Recent osteoarticular pathology (i.e. less than three months) of the lower limbs, whether traumatic or not
* Unfit to consent or refusal to participate in the study
* Obvious standing balance disorder or disabling neurological pathology
* Pain of the musculoskeletal system (joint, tendon or muscle) permanent or during exercise
* Fatigue (evaluation using the Borg scale) during the clinical examination (> 6) prior to performing the sporting gesture
* Known skin allergy to any adhesive product

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Knee abduction moment (quantitative measure) during unplanned sidestep cutting manœuvre. | Inclusion
  The measurement will be the average of the maximum knee abduction moments when the lower extremity is supported on the pushing leg, over the 5 tests carried out with a sidestep cutting manœuvre.

SECONDARY OUTCOMES:
Knee abduction moment when landing jumps in the Single leg Drop Vertical Jump. | Inclusion
  The measurement will be made on the average of the abduction moments of the knee when landing the jump on the ground.
  The subject will perform 3 consecutive jumps in the strictest respect of the instructions.
Star Excursion Balance Test performance. | Inclusion
  The value obtained (in centimeters or relative to the length of the lower limb) reflects the dynamic postural performance of the lower limb under load without specificity of a particular joint of the lower limb. The subject will have 4 training trials per direction on each lower limb then 3 trials will be recorded in order to keep the average.
Angles of ankles, knees, hips, orientation of the pelvis during changes of direction. | Inclusion
  The angles, in degrees, of ankles, knees, hips and orientation of the pelvis during changes of direction will be determined during the unplanned sidestep cutting manœuvre test by computer reconstruction. The values will allow to compare biomechanicals characteristics according to the proprioceptive profile (plastic subjects vs rigid subjects).
Percentage of subjects with a proprioceptive plastic profile. | Inclusion
  A dRPW of 1 indicates 100% use of information from the ankle, while a dRPW of 0 indicates 100% use of information from the hip. It is thus possible to calculate an evolution of this dRPW during the passage from a stable to unstable soil. The "plastic" subjects decreases their dRPW on unstable ground (compared to stable) ("normal" behavior). "Rigid" subjects maintain (or even increase) their dRPW when passing over unstable ground.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REMY-NERIS, Principal Investigator — CHRU BREST
Locations (1):
- CHRU Brest, Brest, France, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Mancini GB, Friedman HZ, Hramiec JE, DeBoe SF. Relation between graded, subcritical impairments of coronary flow reserve and regional myocardial dysfunction induced by isoproterenol infusion in dogs. Am Heart J. 1987 Apr;113(4):906-16. doi: 10.1016/0002-8703(87)90051-2. PMID 3565241
- [Background] Strand T, Tvedte R, Engebretsen L, Tegnander A. [Anterior cruciate ligament injuries in handball playing. Mechanisms and incidence of injuries]. Tidsskr Nor Laegeforen. 1990 Jun 30;110(17):2222-5. Norwegian. PMID 2375011
- [Background] Majewski M, Susanne H, Klaus S. Epidemiology of athletic knee injuries: A 10-year study. Knee. 2006 Jun;13(3):184-8. doi: 10.1016/j.knee.2006.01.005. Epub 2006 Apr 17. PMID 16603363
- [Background] Giroto N, Hespanhol Junior LC, Gomes MR, Lopes AD. Incidence and risk factors of injuries in Brazilian elite handball players: A prospective cohort study. Scand J Med Sci Sports. 2017 Feb;27(2):195-202. doi: 10.1111/sms.12636. Epub 2015 Dec 10. PMID 26661576
- [Background] Olsen OE, Myklebust G, Engebretsen L, Bahr R. Injury mechanisms for anterior cruciate ligament injuries in team handball: a systematic video analysis. Am J Sports Med. 2004 Jun;32(4):1002-12. doi: 10.1177/0363546503261724. PMID 15150050
- [Background] Petersen W, Braun C, Bock W, Schmidt K, Weimann A, Drescher W, Eiling E, Stange R, Fuchs T, Hedderich J, Zantop T. A controlled prospective case control study of a prevention training program in female team handball players: the German experience. Arch Orthop Trauma Surg. 2005 Nov;125(9):614-21. doi: 10.1007/s00402-005-0793-7. PMID 15703919
- [Background] Boden BP, Torg JS, Knowles SB, Hewett TE. Video analysis of anterior cruciate ligament injury: abnormalities in hip and ankle kinematics. Am J Sports Med. 2009 Feb;37(2):252-9. doi: 10.1177/0363546508328107. PMID 19182110
- [Background] Koga H, Nakamae A, Shima Y, Iwasa J, Myklebust G, Engebretsen L, Bahr R, Krosshaug T. Mechanisms for noncontact anterior cruciate ligament injuries: knee joint kinematics in 10 injury situations from female team handball and basketball. Am J Sports Med. 2010 Nov;38(11):2218-25. doi: 10.1177/0363546510373570. Epub 2010 Jul 1. PMID 20595545
- [Background] Krosshaug T, Slauterbeck JR, Engebretsen L, Bahr R. Biomechanical analysis of anterior cruciate ligament injury mechanisms: three-dimensional motion reconstruction from video sequences. Scand J Med Sci Sports. 2007 Oct;17(5):508-19. doi: 10.1111/j.1600-0838.2006.00558.x. Epub 2006 Dec 20. PMID 17181770
- [Background] Prodromos CC, Han Y, Rogowski J, Joyce B, Shi K. A meta-analysis of the incidence of anterior cruciate ligament tears as a function of gender, sport, and a knee injury-reduction regimen. Arthroscopy. 2007 Dec;23(12):1320-1325.e6. doi: 10.1016/j.arthro.2007.07.003. PMID 18063176
- [Background] Rizzo M, Holler SB, Bassett FH 3rd. Comparison of males' and females' ratios of anterior-cruciate-ligament width to femoral-intercondylar-notch width: a cadaveric study. Am J Orthop (Belle Mead NJ). 2001 Aug;30(8):660-4. PMID 11520024
- [Background] Zeng C, Gao SG, Wei J, Yang TB, Cheng L, Luo W, Tu M, Xie Q, Hu Z, Liu PF, Li H, Yang T, Zhou B, Lei GH. The influence of the intercondylar notch dimensions on injury of the anterior cruciate ligament: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2013 Apr;21(4):804-15. doi: 10.1007/s00167-012-2166-4. Epub 2012 Aug 15. PMID 22893267
- [Background] Chaudhari AM, Lindenfeld TN, Andriacchi TP, Hewett TE, Riccobene J, Myer GD, Noyes FR. Knee and hip loading patterns at different phases in the menstrual cycle: implications for the gender difference in anterior cruciate ligament injury rates. Am J Sports Med. 2007 May;35(5):793-800. doi: 10.1177/0363546506297537. Epub 2007 Feb 16. PMID 17307891
- [Background] Hewett TE, Zazulak BT, Myer GD. Effects of the menstrual cycle on anterior cruciate ligament injury risk: a systematic review. Am J Sports Med. 2007 Apr;35(4):659-68. doi: 10.1177/0363546506295699. Epub 2007 Feb 9. PMID 17293469
- [Background] Wojtys EM, Huston LJ, Boynton MD, Spindler KP, Lindenfeld TN. The effect of the menstrual cycle on anterior cruciate ligament injuries in women as determined by hormone levels. Am J Sports Med. 2002 Mar-Apr;30(2):182-8. doi: 10.1177/03635465020300020601. PMID 11912085
- [Background] Hewett TE, Webster KE, Hurd WJ. Systematic Selection of Key Logistic Regression Variables for Risk Prediction Analyses: A Five-Factor Maximum Model. Clin J Sport Med. 2019 Jan;29(1):78-85. doi: 10.1097/JSM.0000000000000486. PMID 28817414
- [Background] Pappas E, Shiyko MP, Ford KR, Myer GD, Hewett TE. Biomechanical Deficit Profiles Associated with ACL Injury Risk in Female Athletes. Med Sci Sports Exerc. 2016 Jan;48(1):107-13. doi: 10.1249/MSS.0000000000000750. PMID 26258858
- [Background] Arundale AJH, Bizzini M, Giordano A, Hewett TE, Logerstedt DS, Mandelbaum B, Scalzitti DA, Silvers-Granelli H, Snyder-Mackler L. Exercise-Based Knee and Anterior Cruciate Ligament Injury Prevention. J Orthop Sports Phys Ther. 2018 Sep;48(9):A1-A42. doi: 10.2519/jospt.2018.0303. PMID 30170521
- [Background] Taylor JB, Waxman JP, Richter SJ, Shultz SJ. Evaluation of the effectiveness of anterior cruciate ligament injury prevention programme training components: a systematic review and meta-analysis. Br J Sports Med. 2015 Jan;49(2):79-87. doi: 10.1136/bjsports-2013-092358. Epub 2013 Aug 6. PMID 23922282
- [Background] Yoo JH, Lim BO, Ha M, Lee SW, Oh SJ, Lee YS, Kim JG. A meta-analysis of the effect of neuromuscular training on the prevention of the anterior cruciate ligament injury in female athletes. Knee Surg Sports Traumatol Arthrosc. 2010 Jun;18(6):824-30. doi: 10.1007/s00167-009-0901-2. Epub 2009 Sep 4. PMID 19760399
- [Background] Grimm NL, Jacobs JC Jr, Kim J, Denney BS, Shea KG. Anterior Cruciate Ligament and Knee Injury Prevention Programs for Soccer Players: A Systematic Review and Meta-analysis. Am J Sports Med. 2015 Aug;43(8):2049-56. doi: 10.1177/0363546514556737. Epub 2014 Dec 1. PMID 25451790
- [Background] Stevenson JH, Beattie CS, Schwartz JB, Busconi BD. Assessing the effectiveness of neuromuscular training programs in reducing the incidence of anterior cruciate ligament injuries in female athletes: a systematic review. Am J Sports Med. 2015 Feb;43(2):482-90. doi: 10.1177/0363546514523388. Epub 2014 Feb 25. PMID 24569703
- [Background] Taylor JB, Ford KR, Schmitz RJ, Ross SE, Ackerman TA, Shultz SJ. Sport-specific biomechanical responses to an ACL injury prevention programme: A randomised controlled trial. J Sports Sci. 2018 Nov;36(21):2492-2501. doi: 10.1080/02640414.2018.1465723. Epub 2018 Apr 19. PMID 29671383
- [Background] Neto T, Sayer T, Theisen D, Mierau A. Functional Brain Plasticity Associated with ACL Injury: A Scoping Review of Current Evidence. Neural Plast. 2019 Dec 27;2019:3480512. doi: 10.1155/2019/3480512. eCollection 2019. PMID 31949428
- [Background] Shultz SJ, Schmitz RJ, Cameron KL, Ford KR, Grooms DR, Lepley LK, Myer GD, Pietrosimone B. Anterior Cruciate Ligament Research Retreat VIII Summary Statement: An Update on Injury Risk Identification and Prevention Across the Anterior Cruciate Ligament Injury Continuum, March 14-16, 2019, Greensboro, NC. J Athl Train. 2019 Sep;54(9):970-984. doi: 10.4085/1062-6050-54.084. Epub 2019 Aug 28. No abstract available. PMID 31461312
- [Background] Fox AS, Bonacci J, McLean SG, Spittle M, Saunders N. What is normal? Female lower limb kinematic profiles during athletic tasks used to examine anterior cruciate ligament injury risk: a systematic review. Sports Med. 2014 Jun;44(6):815-32. doi: 10.1007/s40279-014-0168-8. PMID 24682949
- [Background] Kristianslund E, Faul O, Bahr R, Myklebust G, Krosshaug T. Sidestep cutting technique and knee abduction loading: implications for ACL prevention exercises. Br J Sports Med. 2014 May;48(9):779-83. doi: 10.1136/bjsports-2012-091370. Epub 2012 Dec 20. PMID 23258848
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] Dingenen B, Malfait B, Nijs S, Peers KH, Vereecken S, Verschueren SM, Staes FF. Can two-dimensional video analysis during single-leg drop vertical jumps help identify non-contact knee injury risk? A one-year prospective study. Clin Biomech (Bristol). 2015 Oct;30(8):781-7. doi: 10.1016/j.clinbiomech.2015.06.013. Epub 2015 Jun 26. PMID 26144662
- [Background] Numata H, Nakase J, Kitaoka K, Shima Y, Oshima T, Takata Y, Shimozaki K, Tsuchiya H. Two-dimensional motion analysis of dynamic knee valgus identifies female high school athletes at risk of non-contact anterior cruciate ligament injury. Knee Surg Sports Traumatol Arthrosc. 2018 Feb;26(2):442-447. doi: 10.1007/s00167-017-4681-9. Epub 2017 Aug 24. PMID 28840276
- [Background] Dempsey AR, Lloyd DG, Elliott BC, Steele JR, Munro BJ, Russo KA. The effect of technique change on knee loads during sidestep cutting. Med Sci Sports Exerc. 2007 Oct;39(10):1765-73. doi: 10.1249/mss.0b013e31812f56d1. PMID 17909404
- [Background] Sigward SM, Powers CM. Loading characteristics of females exhibiting excessive valgus moments during cutting. Clin Biomech (Bristol). 2007 Aug;22(7):827-33. doi: 10.1016/j.clinbiomech.2007.04.003. Epub 2007 May 24. PMID 17531364
- [Background] Hewett TE, Myer GD. The mechanistic connection between the trunk, hip, knee, and anterior cruciate ligament injury. Exerc Sport Sci Rev. 2011 Oct;39(4):161-6. doi: 10.1097/JES.0b013e3182297439. PMID 21799427
- [Background] Ford KR, Shapiro R, Myer GD, Van Den Bogert AJ, Hewett TE. Longitudinal sex differences during landing in knee abduction in young athletes. Med Sci Sports Exerc. 2010 Oct;42(10):1923-31. doi: 10.1249/MSS.0b013e3181dc99b1. PMID 20305577
- [Background] Pollard CD, Sigward SM, Powers CM. Limited hip and knee flexion during landing is associated with increased frontal plane knee motion and moments. Clin Biomech (Bristol). 2010 Feb;25(2):142-6. doi: 10.1016/j.clinbiomech.2009.10.005. Epub 2009 Nov 13. PMID 19913961
- [Background] Lawrence RK 3rd, Kernozek TW, Miller EJ, Torry MR, Reuteman P. Influences of hip external rotation strength on knee mechanics during single-leg drop landings in females. Clin Biomech (Bristol). 2008 Jul;23(6):806-13. doi: 10.1016/j.clinbiomech.2008.02.009. Epub 2008 Apr 18. PMID 18395310
- [Background] Nguyen AD, Taylor JB, Wimbish TG, Keith JL, Ford KR. Preferred Hip Strategy During Landing Reduces Knee Abduction Moment in Collegiate Female Soccer Players. J Sport Rehabil. 2018 May 1;27(3):213-217. doi: 10.1123/jsr.2016-0026. Epub 2018 Apr 23. PMID 28338388
- [Background] Sigward SM, Pollard CD, Havens KL, Powers CM. Influence of sex and maturation on knee mechanics during side-step cutting. Med Sci Sports Exerc. 2012 Aug;44(8):1497-503. doi: 10.1249/MSS.0b013e31824e8813. PMID 22330027
- [Background] Stearns KM, Keim RG, Powers CM. Influence of relative hip and knee extensor muscle strength on landing biomechanics. Med Sci Sports Exerc. 2013 May;45(5):935-41. doi: 10.1249/MSS.0b013e31827c0b94. PMID 23190597
- [Background] Zazulak BT, Hewett TE, Reeves NP, Goldberg B, Cholewicki J. Deficits in neuromuscular control of the trunk predict knee injury risk: a prospective biomechanical-epidemiologic study. Am J Sports Med. 2007 Jul;35(7):1123-30. doi: 10.1177/0363546507301585. Epub 2007 Apr 27. PMID 17468378
- [Background] Zazulak BT, Hewett TE, Reeves NP, Goldberg B, Cholewicki J. The effects of core proprioception on knee injury: a prospective biomechanical-epidemiological study. Am J Sports Med. 2007 Mar;35(3):368-73. doi: 10.1177/0363546506297909. Epub 2007 Jan 31. PMID 17267766
- [Background] Decker MJ, Torry MR, Wyland DJ, Sterett WI, Richard Steadman J. Gender differences in lower extremity kinematics, kinetics and energy absorption during landing. Clin Biomech (Bristol). 2003 Aug;18(7):662-9. doi: 10.1016/s0268-0033(03)00090-1. PMID 12880714
- [Background] Hewett TE, Ford KR, Xu YY, Khoury J, Myer GD. Utilization of ACL Injury Biomechanical and Neuromuscular Risk Profile Analysis to Determine the Effectiveness of Neuromuscular Training. Am J Sports Med. 2016 Dec;44(12):3146-3151. doi: 10.1177/0363546516656373. Epub 2016 Jul 29. PMID 27474385
- [Background] Griffin LY, Agel J, Albohm MJ, Arendt EA, Dick RW, Garrett WE, Garrick JG, Hewett TE, Huston L, Ireland ML, Johnson RJ, Kibler WB, Lephart S, Lewis JL, Lindenfeld TN, Mandelbaum BR, Marchak P, Teitz CC, Wojtys EM. Noncontact anterior cruciate ligament injuries: risk factors and prevention strategies. J Am Acad Orthop Surg. 2000 May-Jun;8(3):141-50. doi: 10.5435/00124635-200005000-00001. PMID 10874221
- [Background] Mendiguchia J, Ford KR, Quatman CE, Alentorn-Geli E, Hewett TE. Sex differences in proximal control of the knee joint. Sports Med. 2011 Jul 1;41(7):541-57. doi: 10.2165/11589140-000000000-00000. PMID 21688868
- [Background] Myer GD, Brent JL, Ford KR, Hewett TE. A pilot study to determine the effect of trunk and hip focused neuromuscular training on hip and knee isokinetic strength. Br J Sports Med. 2008 Jul;42(7):614-9. doi: 10.1136/bjsm.2007.046086. Epub 2008 Feb 28. PMID 18308886
- [Background] Bonnette S, Diekfuss JA, Grooms DR, Kiefer AW, Riley MA, Riehm C, Moore C, Barber Foss KD, DiCesare CA, Baumeister J, Myer GD. Electrocortical dynamics differentiate athletes exhibiting low- and high- ACL injury risk biomechanics. Psychophysiology. 2020 Apr;57(4):e13530. doi: 10.1111/psyp.13530. Epub 2020 Jan 20. PMID 31957903
- [Background] Swanik CB. Brains and Sprains: The Brain's Role in Noncontact Anterior Cruciate Ligament Injuries. J Athl Train. 2015 Oct;50(10):1100-2. doi: 10.4085/1062-6050-50.10.08. Epub 2015 Sep 4. PMID 26340611
- [Background] Grooms DR, Page SJ, Nichols-Larsen DS, Chaudhari AM, White SE, Onate JA. Neuroplasticity Associated With Anterior Cruciate Ligament Reconstruction. J Orthop Sports Phys Ther. 2017 Mar;47(3):180-189. doi: 10.2519/jospt.2017.7003. Epub 2016 Nov 5. PMID 27817301
- [Background] Needle AR, Lepley AS, Grooms DR. Central Nervous System Adaptation After Ligamentous Injury: a Summary of Theories, Evidence, and Clinical Interpretation. Sports Med. 2017 Jul;47(7):1271-1288. doi: 10.1007/s40279-016-0666-y. PMID 28005191
- [Background] Swanik CB, Covassin T, Stearne DJ, Schatz P. The relationship between neurocognitive function and noncontact anterior cruciate ligament injuries. Am J Sports Med. 2007 Jun;35(6):943-8. doi: 10.1177/0363546507299532. Epub 2007 Mar 16. PMID 17369562
- [Background] Grindstaff TL, Jackson KR, Garrison JC, Diduch DR, Ingersoll CD. Decreased quadriceps activation measured hours prior to a noncontact anterior cruciate ligament tear. J Orthop Sports Phys Ther. 2008 Aug;38(8):508-16. doi: 10.2519/jospt.2008.2761. Epub 2008 Aug 1. PMID 18678959
- [Background] Diekfuss JA, Grooms DR, Yuan W, Dudley J, Barber Foss KD, Thomas S, Ellis JD, Schneider DK, Leach J, Bonnette S, Myer GD. Does brain functional connectivity contribute to musculoskeletal injury? A preliminary prospective analysis of a neural biomarker of ACL injury risk. J Sci Med Sport. 2019 Feb;22(2):169-174. doi: 10.1016/j.jsams.2018.07.004. Epub 2018 Jul 10. PMID 30017465
- [Background] Diekfuss JA, Grooms DR, Nissen KS, Schneider DK, Foss KDB, Thomas S, Bonnette S, Dudley JA, Yuan W, Reddington DL, Ellis JD, Leach J, Gordon M, Lindsey C, Rushford K, Shafer C, Myer GD. Alterations in knee sensorimotor brain functional connectivity contributes to ACL injury in male high-school football players: a prospective neuroimaging analysis. Braz J Phys Ther. 2020 Sep-Oct;24(5):415-423. doi: 10.1016/j.bjpt.2019.07.004. Epub 2019 Jul 17. PMID 31377125
- [Background] Grooms DR, Page S, Onate JA. Brain Activation for Knee Movement Measured Days Before Second Anterior Cruciate Ligament Injury: Neuroimaging in Musculoskeletal Medicine. J Athl Train. 2015 Sep 29. doi: 10.4085/1062-6050-50-10-02. Online ahead of print. PMID 26418959
- [Background] Goossens N, Janssens L, Caeyenberghs K, Albouy G, Brumagne S. Differences in brain processing of proprioception related to postural control in patients with recurrent non-specific low back pain and healthy controls. Neuroimage Clin. 2019;23:101881. doi: 10.1016/j.nicl.2019.101881. Epub 2019 May 28. PMID 31163385
- [Background] Monjo F, Forestier N. Movement unpredictability and temporal constraints affect the integration of muscle fatigue information into forward models. Neuroscience. 2014 Sep 26;277:584-94. doi: 10.1016/j.neuroscience.2014.07.055. Epub 2014 Jul 30. PMID 25086315
- [Background] Peterka RJ. Sensory integration for human balance control. Handb Clin Neurol. 2018;159:27-42. doi: 10.1016/B978-0-444-63916-5.00002-1. PMID 30482320
- [Background] Vuillerme N, Danion F, Marin L, Boyadjian A, Prieur JM, Weise I, Nougier V. The effect of expertise in gymnastics on postural control. Neurosci Lett. 2001 May 4;303(2):83-6. doi: 10.1016/s0304-3940(01)01722-0. PMID 11311498
- [Background] Grooms DR, Onate JA. Neuroscience Application to Noncontact Anterior Cruciate Ligament Injury Prevention. Sports Health. 2016 Mar-Apr;8(2):149-52. doi: 10.1177/1941738115619164. PMID 26608453
- [Background] Koga H, Nakamae A, Shima Y, Bahr R, Krosshaug T. Hip and Ankle Kinematics in Noncontact Anterior Cruciate Ligament Injury Situations: Video Analysis Using Model-Based Image Matching. Am J Sports Med. 2018 Feb;46(2):333-340. doi: 10.1177/0363546517732750. Epub 2017 Oct 12. PMID 29024605
- [Background] Kiers H, Brumagne S, van Dieen J, Vanhees L. Test-retest reliability of muscle vibration effects on postural sway. Gait Posture. 2014;40(1):166-71. doi: 10.1016/j.gaitpost.2014.03.184. Epub 2014 Apr 3. PMID 24794420
- [Background] Eklund G. General features of vibration-induced effects on balance. Ups J Med Sci. 1972;77(2):112-24. doi: 10.1517/03009734000000016. No abstract available. PMID 4262735
- [Background] Roll JP, Vedel JP. Kinaesthetic role of muscle afferents in man, studied by tendon vibration and microneurography. Exp Brain Res. 1982;47(2):177-90. doi: 10.1007/BF00239377. PMID 6214420
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281
- [Background] Forestier N, Terrier R, Teasdale N. Ankle muscular proprioceptive signals' relevance for balance control on various support surfaces: an exploratory study. Am J Phys Med Rehabil. 2015 Jan;94(1):20-7. doi: 10.1097/PHM.0000000000000137. PMID 24919080
- [Background] Ivanenko YP, Talis VL, Kazennikov OV. Support stability influences postural responses to muscle vibration in humans. Eur J Neurosci. 1999 Feb;11(2):647-54. doi: 10.1046/j.1460-9568.1999.00471.x. PMID 10051765
- [Background] Brumagne S, Cordo P, Verschueren S. Proprioceptive weighting changes in persons with low back pain and elderly persons during upright standing. Neurosci Lett. 2004 Aug 5;366(1):63-6. doi: 10.1016/j.neulet.2004.05.013. PMID 15265591
- [Background] Kiers H, Brumagne S, van Dieen J, van der Wees P, Vanhees L. Ankle proprioception is not targeted by exercises on an unstable surface. Eur J Appl Physiol. 2012 Apr;112(4):1577-85. doi: 10.1007/s00421-011-2124-8. Epub 2011 Aug 21. PMID 21858665
- [Background] Brumagne S, Diers M, Danneels L, Moseley GL, Hodges PW. Neuroplasticity of Sensorimotor Control in Low Back Pain. J Orthop Sports Phys Ther. 2019 Jun;49(6):402-414. doi: 10.2519/jospt.2019.8489. PMID 31151373
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876
- [Background] Lubetzky AV, McCoy SW, Price R, Kartin D. Response to Tendon Vibration Questions the Underlying Rationale of Proprioceptive Training. J Athl Train. 2017 Feb;52(2):97-107. doi: 10.4085/1062-6050-52.1.06. Epub 2017 Jan 26. PMID 28125270
- [Background] Claeys K, Dankaerts W, Janssens L, Pijnenburg M, Goossens N, Brumagne S. Young individuals with a more ankle-steered proprioceptive control strategy may develop mild non-specific low back pain. J Electromyogr Kinesiol. 2015 Apr;25(2):329-38. doi: 10.1016/j.jelekin.2014.10.013. Epub 2014 Oct 31. PMID 25467548
- [Background] Bonnet CT, Lepeut M. Proximal postural control mechanisms may be exaggeratedly adopted by individuals with peripheral deficiencies: a review. J Mot Behav. 2011;43(4):319-28. doi: 10.1080/00222895.2011.589415. Epub 2011 Jul 6. PMID 21732867
- [Background] van den Hoorn W, Kerr GK, van Dieen JH, Hodges PW. Center of Pressure Motion After Calf Vibration Is More Random in Fallers Than Non-fallers: Prospective Study of Older Individuals. Front Physiol. 2018 Mar 26;9:273. doi: 10.3389/fphys.2018.00273. eCollection 2018. PMID 29632494
- [Background] Peterka RJ. Sensorimotor integration in human postural control. J Neurophysiol. 2002 Sep;88(3):1097-118. doi: 10.1152/jn.2002.88.3.1097. PMID 12205132
- [Result] Picot B, Lempereur M, Morel B, Forestier N, Remy-Neris O. Lack of Proprioceptive Strategy Modulation Leads to At-Risk Biomechanics for Anterior Cruciate Ligament in Healthy Athletes. Med Sci Sports Exerc. 2024 May 1;56(5):942-952. doi: 10.1249/MSS.0000000000003378. Epub 2024 Jan 8. PMID 38190373
- See also: Laver L, Landreau P, Seil R, Popovic N, éditeurs. Handball Sports Medicine [Internet]. Berlin, Heidelberg: Springer Berlin Heidelberg; 2018 — http://link.springer.com/10.1007/978-3-662-55892-8
- See also: Laver L, Myklebust G. Handball Injuries: Epidemiology and Injury Characterization. In: Doral MN, Karlsson J, éditeurs. Sports Injuries: Prevention, Diagnosis, Treatment and Rehabilitation — https://doi.org/10.1007/978-3-642-36569-0_287